CLINICAL TRIAL: NCT05574062
Title: Evaluation of the MiniMed 780 System in Young Paediatric Subjects (2-6 Years Old) With Type 1 Diabetes in a Home Setting (LENNY)
Brief Title: Evaluation of the MiniMed 780 System in Paediatric Subjects
Acronym: LENNY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIP342
Record Dates: First submitted 2022-09-22; First posted 2022-10-10 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-04

CONDITIONS: Diabetes type1; Children, Only

STUDY DESIGN:
Intervention Model Description: Run-in Phase: training on the MiniMed 780G system in Manual Mode with SBL activated to collect 2 weeks of baseline data.
  Study Phase:
  Sequence A: subjects MiniMed 780G system in Auto Mode for 12 weeks (Treatment). The washout phase of 2 weeks will be followed by a 12-week phase where subjects will use 780G system in Manual Mode with SBL activated (Control).
  Sequence B: subjects 780G system in Manual Mode with SBL activated (Control). After a washout phase of 2 weeks, subjects will use t MiniMed 780G system in Auto Mode for 12 weeks (Treatment).
  Continuation Phase:
  Period 1: subjects will use MiniMed 780G system in Auto Mode for 18 weeks +/- 6 weeks.
  Period 2:
  Arm A2: subjects will start using the MiniMed 780G BLE 2.0 system (treatment) for 12 weeks (Treatment).
  Arm B2: subjects will continue to use MiniMed™ 780G system in Auto Mode for 12 weeks (Control).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (5):
- All subjects (Other): All subjects used the MiniMed 780G (with G4S sensor) system in Manual Mode for 2 weeks during the run-in phase and used the MiniMed™ 780G system in Auto Mode for 18 weeks during the continuation phase period 1
  Interventions: Device: MiniMed 780G Auto Mode with G4S sensor; Device: MiniMed 780G Manual Mode with G4S sensor
- Study phase - Sequence A (Experimental): Subjects used the MiniMed 780G (with G4S sensor) system in Auto Mode for 12 weeks (Treatment), followed by 2 weeks of washout period where the system was used in Manual Mode with SBL activated (Control).
  After the washout period the subjects used the MiniMed 780G (with G4S sensor) system in Manual Mode with SBL activated (Control).
  Interventions: Device: MiniMed 780G Auto Mode with G4S sensor; Device: MiniMed 780G Manual Mode with G4S sensor
- Study phase - Sequence B (Experimental): Subjects used the MiniMed 780G (with G4S sensor) system in Manual Mode with SBL activated for 12 weeks (Control), followed by 2 weeks of washout period where the system was used in Manual Mode with SBL activated (Control).
  After the washout period the subjects used the MiniMed 780G (with G4S sensor) system in Auto Mode (Treatment).
  Interventions: Device: MiniMed 780G Auto Mode with G4S sensor; Device: MiniMed 780G Manual Mode with G4S sensor
- Continuation Phase - Arm A2 (Experimental): Subjects will start using the MiniMed™ 780G BLE 2.0 system in Auto Mode with the DS5 sensor
  Interventions: Device: MiniMed 780G Auto Mode with DS5 sensor
- Continuation Phase - Arm B2 (Active Comparator): Subjects will continue to use MiniMed™ 780G system in Auto Mode with G4S sensor for 12 weeks
  Interventions: Device: MiniMed 780G Auto Mode with G4S sensor

INTERVENTIONS:
Device: MiniMed 780G Auto Mode with G4S sensor — MiniMed™ 780G system in Auto Mode with G4S sensor.
  Arms: All subjects; Continuation Phase - Arm B2; Study phase - Sequence A; Study phase - Sequence B
Device: MiniMed 780G Manual Mode with G4S sensor — MiniMed™ 780G system in Manual Mode.
  Arms: All subjects; Study phase - Sequence A; Study phase - Sequence B
Device: MiniMed 780G Auto Mode with DS5 sensor — MiniMed 780G Auto Mode with DS5 sensor
  Arms: Continuation Phase - Arm A2

SUMMARY:
The purpose of this study is to demonstrate the safety and performance of the MiniMed™ 780G system in pediatric subjects (2-6 years old) with type 1 diabetes in a home setting.

The objective of this study is to evaluate the safety and performance of the MiniMed™ 780G system in Auto Mode firstly in comparison to the MiniMed™ 780G system in Manual Mode with Suspend before low activated (currently available standard therapy) and secondly in comparison to the new MiniMed™ 780G BLE 2.0 system with DS5 sensor in Auto Mode among pediatric population (2-6 years old).

DETAILED DESCRIPTION:
CIP342 study is a pre-market, prospective, open-label, multi-center, randomized crossover trial in paediatric subjects (2-6 years old) with type 1 diabetes. The study consists of a run-in phase, a study phase and a continuation phase.

Run-in Phase:

The purpose of the run-in phase (2 to 4 weeks) is to train subject's parent(s)/legal guardian(s) on the MiniMed 780G system in Manual Mode with Suspend before low (SBL) activated and to collect 2 weeks of baseline data. At the end of Run-in Phase, subjects will be randomized into one of two sequences (A or B).

The MiniMed 780G system is composed by the MiniMed 780G pump used with Guardian 4 Sensor (G4S) and Guardian Transmitter 4.

Study Phase:

* Sequence A: subjects will use the Advanced Hybrid Closed Loop (AHCL) therapy (MiniMed 780G system in Auto Mode) for 12 weeks (Treatment). The washout phase of 2 weeks will be followed by a 12-week phase where subjects will use predictive low-glucose suspend (780G system in Manual Mode with SBL activated) (Control).
* Sequence B: subjects will continue to use predictive low-glucose suspend (MiniMed 780G system in Manual Mode with SBL activated) (Control). After a washout phase of 2 weeks, subjects will use Advanced Hybrid Closed Loop (AHCL) therapy (MiniMed 780G system in Auto Mode) for 12 weeks (Treatment).

During washout period all the subjects will use MiniMed 780G system in Manual Mode with SBL activated.

At the end of Study Phase, subjects will start Continuation Phase that is divided in two periods.

Continuation Phase:

* Period 1: enrolled subjects will enter the continuation phase period 1 and will use MiniMed 780G system in Auto Mode for 18 weeks +/- 6 weeks.
* Period 2: At the end of the continuation phase period 1, subjects will be randomized into 2 arms (A2 and B2). This second randomization is completely independent from the first one in the Study Phase.

Arm A2: Subjects will start using the MiniMed 780G BLE 2.0 system (treatment) for 12 weeks. The MiniMed 780G BLE 2.0 system is composed by the MiniMed 780 BLE 2.0 and Disposable Sensor labeled (DS5)

Arm B2: Subjects will continue to use MiniMed™ 780G system in Auto Mode for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 2 - 6 years at time of screening
2. Has a clinical diagnosis of type 1 diabetes for ≥ 6 months prior to screening as determined via medical record or source documentation by an individual qualified to make a medical diagnosis
3. Is on MDI therapy or CSII with or without CGM prior to screening
4. Has a glycosylated hemoglobin (HbA1c) < 11% (97 mmol/mol) at time of screening visit as processed by a Local Lab
5. Is using or willing to switch to one of the following commercialized available insulins: Humalog (insulin lispro injection) and NovoLog (insulin aspart).
6. Must have a minimum daily insulin requirement (Total Daily Dose) of ≥ 6 units
7. Parent(s)/legal guardian(s) willing to upload data from the pump system, must have Internet access, a compatible computer or mobile phone that meets the requirements for uploading the study pump data at home.
8. Is living with one or more parent(s)/legal guardian(s) knowledgeable about emergency procedures for severe hypoglycemia and able to contact emergency services and study staff.
9. Investigator has confidence that the parent(s)/legal guardian(s) can successfully operate all study devices and is capable of adhering to the protocol
10. Subject and parent(s)/legal guardian(s) willingness to participate in all training sessions as directed by study staff.
11. Subject's parent/legal guardian must be willing and able to provide written informed consent.

Exclusion Criteria:

1. Has Addison's disease, growth hormone deficiency, coeliac disease, hypopituitarism or definite gastroparesis, untreated thyroid disorder, or poorly controlled asthma, per investigator judgment.
2. Is using any anti-diabetic medication other than insulin at the time of screening or plan of using during the study (e.g. pramlintide, DPP-4 inhibitor, GLP-1, agonists/mimetics, metformin, SGLT2 inhibitors).
3. Has taken any oral, injectable, or intravenous (IV) glucocorticoids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV glucocorticoids during the course of the study.
4. Has had renal failure defined by creatinine clearance <30 ml/min, as assessed by local lab test ≤6 months before screening or performed at screening at local lab, as defined by the creatinine-based Cockcroft, CKD-EPI or MDRD equations.
5. Has any unresolved adverse skin conditions in the area of sensor placement (e.g. psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).
6. Is under Control IQ or CamAPS FX or other advanced hybrid closed loop therapy (e.g. DIY, MiniMed 780G) in the previous 3 months before enrollment. Note: For the continuation phase only, subjects using MiniMed 780G can be enrolled.
7. Is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or device in the last 2 weeks before enrollment into this study, as per investigator judgment.
8. Has any other disease or condition that may preclude the patient from participating in the study, per investigator judgment.
9. History of >1 DKA event not related to illness or initial diagnosis in the last 3 months.
10. Parent(s)/legal guardian(s) are part of research staff involved with the study.
11. Parent(s)/legal guardian(s) are illiterate

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Cohen, MD, Study Chair — Medtronic
Locations (12):
- Finland (3):
  - HUS, Espoo
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Italy (4):
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti Ancona, "G. Salesi", Ancona
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli, Napoli
  - Ospedale Maggiore della Carità di Novara, Novara
  - Ospedale Pediatrico Bambino Gesù, Roma
- University Medical Center Ljubljana (UMCL), Ljubljana, Slovenia
- United Kingdom (4):
  - Noah's Ark Children's Hospital for Wales, Cardiff
  - LEEDS TEACHING HOSPITALS NHS TRUST - St James, Leeds
  - Leicester Royal Infirmary, Leicester
  - UCLH (University College London Hospitals), London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Battelino T, Kuusela S, Shetty A, Rabbone I, Cherubini V, Campbell F, Ahomaki R, Tuomaala AK, Peters C, Iafusco D, Sundaram P, Schiaffini R, Cellot J, Gulotta F, Di Piazza F, Cohen O; LENNY study group. Efficacy and safety of automated insulin delivery in children aged 2-6 years (LENNY): an open-label, multicentre, randomised, crossover trial. Lancet Diabetes Endocrinol. 2025 Aug;13(8):662-673. doi: 10.1016/S2213-8587(25)00091-9. Epub 2025 Jun 19. PMID 40544853

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 101 subjects signed the informed consent and were assessed for enrollment. Out of them, 3 screening failures due to the following inclusion criteria not met: "Investigator has confidence that the parent(s)/ legal guardian(s) can successfully operate all study devices and is capable of adhering to the protocol" discontinued the study before starting the run-in phase.
Pre-assignment Details: Run-in period
Groups:
- All Subjects: The entire study population (this group is intended for clarification and reporting into the CT.gov PRS
- Sequence A: Subjects used the MiniMed 780G (with G4S sensor) system in Auto Mode for 12 weeks followed by 2 weeks of washout period where the system was used in Manual Mode with SBL activated. After the washout period the subjects used the MiniMed 780G system in Manual Mode with SBL activated for the remaining 12 weeks.
- Sequence B: Subjects used the MiniMed 780G (with G4S sensor) system in Manual Mode with SBL activated (Sequence B) for 12 weeks followed by 2 weeks of washout period where the system was used in Manual Mode with SBL activated. After the washout period the subjects used the MiniMed 780G system in Auto Mode for the remaining 12 weeks.
- Arm A2: Arm A2: Subjects will start using the MiniMed™ 780G BLE 2.0 system with the DS5 sensor for 12 weeks
- Arm B2: Arm B2: Subjects will continue to use MiniMed™ 780G system in Auto Mode for 12 weeks
Period: Pre Run-In
Arm/Group | All Subjects | Sequence A | Sequence B | Arm A2 | Arm B2
Started | 101 | 0 | 0 | 0 | 0
Completed | 98 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0
Not completed — Screening failure | 3 | 0 | 0 | 0 | 0
Period: Run-in
Arm/Group | All Subjects | Sequence A | Sequence B | Arm A2 | Arm B2
Started | 98 | 0 | 0 | 0 | 0
Completed | 98 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Study Phase Period 1
Arm/Group | All Subjects | Sequence A | Sequence B | Arm A2 | Arm B2
Started | 0 | 50 | 48 | 0 | 0
Completed | 0 | 49 | 48 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Period: Wash-out Period
Arm/Group | All Subjects | Sequence A | Sequence B | Arm A2 | Arm B2
Started | 0 | 49 | 48 | 0 | 0
Completed | 0 | 49 | 48 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Study Phase Period 2
Arm/Group | All Subjects | Sequence A | Sequence B | Arm A2 | Arm B2
Started | 0 | 49 | 48 | 0 | 0
Completed | 0 | 48 | 48 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Period: Continuation Phase Period 1
Arm/Group | All Subjects | Sequence A | Sequence B | Arm A2 | Arm B2
Started | 95 | 0 | 0 | 0 | 0
Completed | 91 | 0 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Period: Continuation Phase Period 2
Arm/Group | All Subjects | Sequence A | Sequence B | Arm A2 | Arm B2
Started | 0 | 0 | 0 | 45 | 46
Completed | 0 | 0 | 0 | 44 | 46
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Phase - Sequence A: Subjects used the MiniMed 780G (with G4S sensor) system in Auto Mode for 12 weeks (Treatment), followed by 2 weeks of washout period where the system was used in Manual Mode with SBL activated (Control).
  After the washout period the subjects used the MiniMed 780G (with G4S sensor) system in Manual Mode with SBL activated (Control).
  MiniMed 780G Auto Mode with G4S sensor: MiniMed™ 780G system in Auto Mode with G4S sensor.
  MiniMed 780G Manual Mode with G4S sensor: MiniMed™ 780G system in Manual Mode.
- Study Phase - Sequence B: Subjects used the MiniMed 780G (with G4S sensor) system in Manual Mode with SBL activated for 12 weeks (Control), followed by 2 weeks of washout period where the system was used in Manual Mode with SBL activated (Control).
  After the washout period the subjects used the MiniMed 780G (with G4S sensor) system in Auto Mode (Treatment).
  MiniMed 780G Auto Mode with G4S sensor: MiniMed™ 780G system in Auto Mode with G4S sensor.
  MiniMed 780G Manual Mode with G4S sensor: MiniMed™ 780G system in Manual Mode.
- Total: Total of all reporting groups
Arm/Group | Study Phase - Sequence A | Study Phase - Sequence B | Total
Number analyzed (Participants) | 50 | 48 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.61 (1.076) | 4.84 (1.234) | 4.72 (1.156)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 27 | 23 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Finland | 12 | 15 | 27
  United Kingdom | 15 | 11 | 26
  Italy | 13 | 12 | 25
  Slovenia | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Study Phase Primary Endpoint: Percentage of Time in Range (TIR 70 to 180 mg/dL [3.9-10.0 mmol/L]) - Non-inferiority Test
Description: The primary endpoint is the between-treatment difference in the percentage of time that the sensor glucose measurement is in the target range, 70 to 180 mg/dL (3.9-10.0 mmol/L), non-inferiority test.
Time Frame: 12 weeks for each cross-over period
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- MiniMed 780G (With G4S Sensor) System in Auto Mode: Data from period 1 for subjects randomized in Sequence A Data from period 2 for subjects randomized in Sequence B
- MiniMed 780G (With G4S Sensor) System in Manual Mode + SBL: Data from period 2 for subjects randomized in Sequence A Data from period 1 for subjects randomized in Sequence B
Arm/Group | MiniMed 780G (With G4S Sensor) System in Auto Mode | MiniMed 780G (With G4S Sensor) System in Manual Mode + SBL
Number analyzed (Participants) | 97 | 97
percentage of time | 68.34 (6.922) | 58.34 (12.455)
Statistical Analysis 1: Comparison: MiniMed 780G (With G4S Sensor) System in Auto Mode vs MiniMed 780G (With G4S Sensor) System in Manual Mode + SBL; Test type: Non-Inferiority — -7.5% non-inferiority margin; Mixed Models Analysis; Mean Difference (Final Values) = 9.88, 95% CI 2-sided [8.04 to 11.72] — Mixed model adjusted for baseline (run-in) values

2. Primary Outcome: Continuation Phase Primary Endpoint: Mean HbA1c (%) - Non-inferiority Test
Description: The primary endpoint for continuation phase is the between-treatment difference in the mean HbA1c (%) at the end of 12-week continuation phase period 2. The endpoint will be assessed for non-inferiority with an absolute margin of 0.4% HbA1c.
Time Frame: The outcome was measured at the end of the 12-week continuation phase period 2
Population: The number of subjects with endpoint measurements available at the end of the continuation phase period 2 were 38 out of 45 and 42 out of 46 for arm A2 and arm B2, respectively
Measure: Mean (Standard Deviation); unit: % of hba1c
Groups:
- MiniMed™ 780G System in Auto Mode With the DS5 Sensor: Subjects used the MiniMed™ 780G system in auto mode with the DS5 sensor for 12 weeks during the continuation phase period 2
- MiniMed™ 780G System in Auto Mode With the G4S Sensor: Subjects used the MiniMed™ 780G system in auto mode with the G4S sensor for 12 weeks during the continuation phase period 2
Arm/Group | MiniMed™ 780G System in Auto Mode With the DS5 Sensor | MiniMed™ 780G System in Auto Mode With the G4S Sensor
Number analyzed (Participants) | 38 | 42
% of hba1c | 7.30 (0.529) | 7.24 (0.643)
Statistical Analysis 1: Comparison: MiniMed™ 780G System in Auto Mode With the DS5 Sensor vs MiniMed™ 780G System in Auto Mode With the G4S Sensor; Test type: Non-Inferiority — non-inferiority margin of 0.4% HbA1c; Regression, Linear; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.03 to 0.31] — Linear regression model adjusted for baseline (continuation phase period1) values

3. Secondary Outcome: Study Phase Secondary Endpoint 1- Mean HbA1c (%) - Non-inferiority Test
Description: Between-treatment difference in mean HbA1c at the end of each 12-week cross-over period, non-inferiority test.
Time Frame: The outcome was measured at the end of each 12 week cross-over period
Measure: Mean (Standard Deviation); unit: % of hba1c
Groups:
- MiniMed 78G (With G4S Sensor) System in Manual Mode + SBL: Data from period 2 for subjects randomized in Sequence A Data from period 1 for subjects randomized in Sequence B
Arm/Group | MiniMed 780G (With G4S Sensor) System in Auto Mode | MiniMed 78G (With G4S Sensor) System in Manual Mode + SBL
Number analyzed (Participants) | 97 | 96
% of hba1c | 7.00 (0.533) | 7.61 (0.906)
Statistical Analysis 1: Comparison: MiniMed 780G (With G4S Sensor) System in Auto Mode vs MiniMed 78G (With G4S Sensor) System in Manual Mode + SBL; Test type: Non-Inferiority — non- inferiority margin of 0.4%; Mixed Models Analysis; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.76 to -0.46] — Mixed model adjusted for baseline (screening) values

4. Secondary Outcome: Study Phase Secondary Endpoint 2 - Percentage of Time in Range (TIR 70 to 180 mg/dL [3.9-10.0 mmol/L]) - Superiority Test
Description: Between-treatment difference in % Time spent in target range (70 to 180 mg/dL [3.9-10.0 mmol/L]), during each 12 week cross-over period, superiority test.
Time Frame: 12 weeks for each cross-over period
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | MiniMed 780G (With G4S Sensor) System in Auto Mode | MiniMed 78G (With G4S Sensor) System in Manual Mode + SBL
Number analyzed (Participants) | 97 | 97
percentage of time | 68.34 (6.922) | 58.34 (12.455)
Statistical Analysis 1: Comparison: MiniMed 780G (With G4S Sensor) System in Auto Mode vs MiniMed 78G (With G4S Sensor) System in Manual Mode + SBL; Test type: Superiority; p < .0001, Mixed Models Analysis; Median Difference (Final Values) = 9.88, 95% CI 2-sided [8.04 to 11.72] — Mixed model adjusted for baseline (run-in) values

5. Secondary Outcome: Study Phase Secondary Endpoint 3 - Mean HbA1c (%) - Superiority Test.
Description: Between-treatment difference in mean HbA1c at the end of each 12-week cross-over period, superiority test.
Time Frame: The outcome was measured at the end of each 12 week cross-over period
Measure: Mean (Standard Deviation); unit: % of hba1c
Arm/Group | MiniMed 780G (With G4S Sensor) System in Auto Mode | MiniMed 78G (With G4S Sensor) System in Manual Mode + SBL
Number analyzed (Participants) | 97 | 96
% of hba1c | 7.00 (0.533) | 7.61 (0.906)
Statistical Analysis 1: Comparison: MiniMed 780G (With G4S Sensor) System in Auto Mode vs MiniMed 78G (With G4S Sensor) System in Manual Mode + SBL; Test type: Superiority; p < .0001, Mixed Models Analysis; Mean Difference (Net) = -0.61, 95% CI 2-sided [-0.76 to -0.46] — Mixed model adjusted for baseline (screening) values

6. Secondary Outcome: Continuation Phase Secondary Endpoint 1- Mean HbA1c (%) - Superiority Test
Description: Between-treatment difference in Mean HbA1c at the end of the 12-week continuation phase period 2, superiority test.
Time Frame: The outcome was measured at the end of the 12-week continuation phase period 2
Measure: Mean (Standard Deviation); unit: % of hba1c
Groups:
- MiniMed™ 780G System in Auto Mode With the G4S: Subjects used the MiniMed™ 780G system in auto mode with the G4S sensor for 12 weeks during the continuation phase period 2
Arm/Group | MiniMed™ 780G System in Auto Mode With the DS5 Sensor | MiniMed™ 780G System in Auto Mode With the G4S
Number analyzed (Participants) | 38 | 42
% of hba1c | 7.30 (0.529) | 7.24 (0.643)
Statistical Analysis 1: Comparison: MiniMed™ 780G System in Auto Mode With the DS5 Sensor vs MiniMed™ 780G System in Auto Mode With the G4S; Test type: Superiority; p = 0.1097, Regression, Linear; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.03 to 0.31] — Linear regression model adjusted for baseline (period1) values

7. Secondary Outcome: Continuation Phase Secondary Endpoint 2- Percentage of Time in Range (TIR 70 to 180 mg/dL [3.9-10.0 mmol/L]) - Non-inferiority Test
Description: Between-treatment difference in % Time spent in target range (70 to 180 mg/dL [3.9-10.0 mmol/L]) during the end 12-week continuation phase period 2, non-inferiority test
Time Frame: 12 weeks of continuation phase period 2
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | MiniMed™ 780G System in Auto Mode With the DS5 Sensor | MiniMed™ 780G System in Auto Mode With the G4S
Number analyzed (Participants) | 44 | 46
percentage of time | 69.7 (7.728) | 68.8 (8.615)
Statistical Analysis 1: Comparison: MiniMed™ 780G System in Auto Mode With the DS5 Sensor vs MiniMed™ 780G System in Auto Mode With the G4S; Test type: Non-Inferiority — non inferiority margin of -7.5%; Regression, Linear; Mean Difference (Net) = 1.17, 95% CI 2-sided [-0.04 to 2.38] — Linear regression adjusted for baseline (continuation phase period 1) values

8. Secondary Outcome: Continuation Phase Secondary Endpoint 3- Percentage of Time in Range (TIR 70 to 180 mg/dL [3.9-10.0 mmol/L]) - Superiority Test
Description: Between-treatment difference in % Time spent in target range (70 to 180 mg/dL [3.9-10.0 mmol/L]) during the end 12-week continuation phase period 2, superiority test.
Time Frame: 12 weeks of continuation phase period 2
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | MiniMed™ 780G System in Auto Mode With the DS5 Sensor | MiniMed™ 780G System in Auto Mode With the G4S
Number analyzed (Participants) | 44 | 46
percentage of time | 69.66 (7.734) | 68.86 (8.615)
Statistical Analysis 1: Comparison: MiniMed™ 780G System in Auto Mode With the DS5 Sensor vs MiniMed™ 780G System in Auto Mode With the G4S; Test type: Superiority; p = 0.0581, Regression, Linear; Mean Difference (Final Values) = 1.17, 95% CI 2-sided [-0.04 to 2.38] — Linear regression adjusted for baseline (continuation phase period 1) values

ADVERSE EVENTS:
Time Frame: AE data were collected from the signature of the informed consent to the end of the continuation phase for approximately 58 weeks (2 weeks of run-in, 12 weeks of period 1, 2 weeks of wash-out, 12 weeks of period 2, 18 weeks of continuation phase period 1 and 12 weeks of continuation phase period 2).
Groups:
- Run-In Period: All Enrolled subjects had a 2 week run-in period before randomization using the MiniMed 780G (with G4S sensor) system in Manual Mode + SBL
- MiniMed 780G (With G4S Sensor) System in Auto Mode - Study Phase: Data from period 1 for subjects randomized in Sequence A Data from period 2 for subjects randomized in Sequence B
- Wash-out Period: 2 week run-in period between cross-over period 1 and period 2 using the MiniMed 780G (with G4S sensor) system in Manual Mode + SBL
- MiniMed 780G (With G4S Sensor) System in Manual Mode + SBL - Study Phase: Data from period 2 for subjects randomized in Sequence A Data from period 1 for subjects randomized in Sequence B
- Continuation Phase Period 1: 18 week period using the MiniMed 780G (with G4S sensor) system in Auto Mode before second randomization
- MiniMed 780G (With DS5 Sensor) System in Auto Mode - Continuation Phase Period 2; MiniMed 780G (With G4S Sensor) System in Auto Mode - Continuation Phase Period 2: Data from continuation phase period 2 for subjects randomized in Arm A2
Arm/Group | Run-In Period | MiniMed 780G (With G4S Sensor) System in Auto Mode - Study Phase | Wash-out Period | MiniMed 780G (With G4S Sensor) System in Manual Mode + SBL - Study Phase | Continuation Phase Period 1 | MiniMed 780G (With DS5 Sensor) System in Auto Mode - Continuation Phase Period 2 | MiniMed 780G (With G4S Sensor) System in Auto Mode - Continuation Phase Period 2
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/98 | 0/97 | 0/97 | 1/95 | 0/45 | 0/46
Serious Adverse Events (participants affected / at risk) | 1/98 | 5/98 | 1/97 | 2/97 | 4/95 | 1/45 | 2/46
Other Adverse Events (participants affected / at risk) | 18/98 | 45/98 | 11/97 | 39/97 | 37/95 | 11/45 | 17/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-In Period (N=98) | MiniMed 780G (With G4S Sensor) System in Auto Mode - Study Phase (N=98) | Wash-out Period (N=97) | MiniMed 780G (With G4S Sensor) System in Manual Mode + SBL - Study Phase (N=97) | Continuation Phase Period 1 (N=95) | MiniMed 780G (With DS5 Sensor) System in Auto Mode - Continuation Phase Period 2 (N=45) | MiniMed 780G (With G4S Sensor) System in Auto Mode - Continuation Phase Period 2 (N=46)
Left tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DKA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral Induced Wheeze (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scarlet Fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower Respiratory Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella infection with secondary supra-infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALLERGIC REACTION TO AMOXICILLIN SUSP (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reactive airway disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MENINGOENCEPHALI TIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-In Period (N=98) | MiniMed 780G (With G4S Sensor) System in Auto Mode - Study Phase (N=98) | Wash-out Period (N=97) | MiniMed 780G (With G4S Sensor) System in Manual Mode + SBL - Study Phase (N=97) | Continuation Phase Period 1 (N=95) | MiniMed 780G (With DS5 Sensor) System in Auto Mode - Continuation Phase Period 2 (N=45) | MiniMed 780G (With G4S Sensor) System in Auto Mode - Continuation Phase Period 2 (N=46)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2) | 6 (7) | 2 (2) | 1 (1) | 7 (7) | 1 (1) | 2 (3)
General disorders and administration site conditions (General disorders) | 10 (10) | 13 (18) | 3 (3) | 9 (12) | 8 (10) | 2 (5) | 4 (4)
Infections and infestations (Infections and infestations) | 6 (6) | 27 (36) | 7 (7) | 31 (48) | 31 (53) | 7 (9) | 11 (18)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 0 (0) | 3 (3) | 3 (3) | 2 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT05574062/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT05574062/SAP_001.pdf